CLINICAL TRIAL: NCT00459303
Title: Intraidivisual Comparison of Functional Vision Provided by AMO Tecnis Z9000 and ALcon SA60AT Acrysof Posterior Chamber Intraocular Lenses
Brief Title: Comparison of Functional Vision Provided by AMO Tecnis Z9000 and Alcon SA60AT Acrysof
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 05012006
Record Dates: First submitted 2007-04-10; First posted 2007-04-11 (Estimated); Results first posted 2014-02-17 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2013-12

CONDITIONS: Cataract
Keywords: cataract; aspherical intraocular lenses; functional vision
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- intraocular lens (Active Comparator): patients with bilateral clinical significant cataract reisiceved cataract surgeries and recieved spherial intraocuar lens(SA60AT, Alcon) in one eye and aspherical intraocular lens(Tecnis Z9000, AMO)in the other respectively.
  Interventions: Device: aspherical intraocular lens; Device: spherical intraocular lens

INTERVENTIONS:
Device: aspherical intraocular lens — implantation of aspherical intraocular lenses(AMO Tecnis Z9000)during cataract suregry (small cornea incision phacoemulsification, deliver with Monarch II device, in the bag implantation)
  Other Names: AMO Tecnis Z9000
Device: spherical intraocular lens — implantation of spherical intraocular lenses(Alcon SA60AT Acrysof)during cataract suregry (small cornea incision phacoemulsification, deliver with Monarch II device, in the bag implantation)
  Other Names: Alcon SA60AT Acrysof

SUMMARY:
This study is to compare intraindividually the functional vision provided by two different posterior chamber intraocular lenses: AMO Tecnis Z9000 and Alcon SA60AT Acrysoft. To see if the aspherical intraocular lenses provide better functional vision than traditional spherical intraocular lenses.

DETAILED DESCRIPTION:
In this prospective study, 20 patients with bilateral catarct presenting for cataract surgery are randomly assigned to recieve an aspherical intraocular lens(AMO Tecnis Z9000) in one eye and a spherical intraocular lens(Alcon SA60AT Acrysof)in the other. All surgeries are performed by one experienced surgeon(Fung-Rong Hu,MD)with clear cornea small incision phacoemulsification and in-the-bag posterior chamber intraocular implantation.

The patients are followed for 3 months, and postoperative contrast sensitivity, contrast acuity, corneal & total ocular high-ordered aberrations are measured and compared intraidividually between two different IOL groups.

Outcome Measurement:

1. Contrast sensitivity testing: measured with spectacle correction for the target distance of three meters using wall-mounted FACT sine-wave grating chart with nine levels of contrast.The graphic contrast sensitivity is recorded as a log functional units on the y-axis and displayed for five spatial frequency targets (1.5, 3, 6, 12, 18 cycles per degree (cpd))on x- axis.
2. Contrast acuity testing: measured with spectacle correction for the target distance of three meters using logMAR letter chart(Precision Vision®)represented on a wall-mounted illuminator cabinet.Two types of contrast charts are used, high contrast(Cat.No.2103 SLOAN translucent chart)and low contrast(Cat.No.2132 10% SLOAN translucent chart),and are tested under both photopic and mesopic conditions.
3. Pupil diameters: measured by Colvard infrared pupillometer (Oasis. Medical, Glendora, CA, USA )under both photopic and mesopic luminance levels.
4. Corneal aberration analysis: performed with TMS-4 (Tomey, Japan).The corneal HOAs are described with Zernike polynomials of 3rd-to 5th- order root-mean-square(RMS)of central 6mm diameter using VOLPro 6.89 software(Fa. Sarver and Associates, Carbondale. Ill, USA).
5. Total ocular aberration analysis: performed with a Hartmann-Shack aberrometer(Zywave, Bausch & Lomb Inc., Rochester, New. York)under maximal mydriasis with Mydrin-P(phenylephrine hydrochloride 0.5% and tropicamide 0.5%, Santen).The wavefront errors were described using Zernike polynomials RMS for total HOA at pupil diameter of 5 mm and 6 mm, primary spherical (Z 4,0) and 3rd-to 5th-order aberration at pupil diameter of 6 mm.

Data Analysis:

* Mann-Whitney U matched-paired test was used with STATA software
* P values of 0.05 or less were considered statistically significant

ELIGIBILITY:
Inclusion Criteria:

* Bilateral cataracts, eligible for phacoemulsification with primary implantation of a posterior chamber IOL
* Willing and able to comply with scheduled visits and other study procedures

Exclusion Criteria:

* Preoperative ocular pathology potentially affect visual acuity. EX: diabetic retinopathy, macular degeneration, corneal opacity, glaucoma, visual field defect...etc.
* Previous ocular surgery. Ex: refractive surgery, vitreoretinal surgery...etc.
* Patients who cannot cooperative with the study procedures

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-10; Primary Completion 2007-09 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Yuang Su, MD, Principal Investigator — National Taiwan Unoversity Hospital; Fung-Rong Hu, MD, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with clinically significant cataract received cataract surgery and implantation of aspherical IOL in one eye and spherical IOL in the contralateral eye. All cases were enrolled from October 2005 to April 2006 and were followed up for at least three months at the department of ophthalmology.
Pre-assignment Details: Patients with diabetes or other systemic disease, such as dysthyroid related orbitopathy or drug related optic neuropathy, that may potentially affect contrast sensitivity and visual quality were excluded.
Groups:
- Cataract Patients: Patients with clinically significant cataract received cataract surgery and implantation of aspherical IOL in one eye and spherical IOL in the contralateral eye.
Period: Overall Study
Arm/Group | Cataract Patients
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cataract Patients
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.4 (9.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Region of Enrollment [Number; unit: participants]
  Taiwan | 20

OUTCOME MEASURES:

1. Primary Outcome: Best Corrected logMAR Contrast Acuity at Photopic/Mesopic Condition
Description: Contrast acuity testing was measured with spectacle correction for the target distance of three meters using a logMAR letter chart (Precision Vision®) represented on a wall-mounted illuminator cabinet. Two types of contrast charts were used, high contrast (Cat.No.2103 SLOAN translucent chart) and low contrast (Cat.No.2132 10% SLOAN translucent chart), and these were tested under both photopic (250 Lux) and mesopic (0.5 Lux) conditions. The contrast acuity tested ranges from 20/160 to 20/20(from worse to best), which equals LogMAR(Logarithm of the Minimum Angle of Resolution)0.9 to -0.3. All of the visual acuity and functional vision testing examinations mentioned above were performed by a single ophthalmologist. The outcomes were recorded as average of three post-operative measurments.
Time Frame: average data of post-op 3rd, 6th, 12th week measurements
Population: we obtained data and calculated the probable sample size needed from the following reference papers:
  1. Ophthalmologe 2005 Jan;102(1):51-7.
  2. Acta Ophthalmol Scand 2004;82(6):718-22.
Measure: Mean (Standard Deviation); unit: log MAR
Groups:
- Spherical Intraocular Lens: patients recieved cataract surgery and recived spherical intraocuar lens(SA60AT, Alcon) in one eye.
- Aspherical Intraocular Lens: patients recieved cataract surgery and recived aspherical intraocuar lens(Tecnis Z9000, AMO) in the other eye.
Arm/Group | Spherical Intraocular Lens | Aspherical Intraocular Lens
Number analyzed (Participants) | 20 | 20
log MAR | 0.34 (0.10) | 0.34 (0.10)

2. Secondary Outcome: Corneal High-order Aberrations
Description: Corneal topography was performed with a TMS-4 corneal tomographer (Tomey, Japan). We used the 31-rings placido-based system that covers 10.9 mm of corneal diameter which is sufficient for the study of aberrations up to the fifth order for 6 mm diameter. Corneal HOAs were described with Zernike polynomials of 3rd- to 5th-order root-mean-square (RMS) of central 6mm diameter using VOLPro 6.89 software (Fa. Sarver and Associates, Carbondale. Ill, USA).
Time Frame: pre-op & averate data of post-op 3rd, 6th, 12th week measurements
Measure: Mean (Standard Deviation); unit: μm
Groups:
- Aspherical Intraocular Lens: patients recieved cataract surgery and recived spherical intraocuar lens(Tecnis Z9000,AMO) in the other eye.
Arm/Group | Spherical Intraocular Lens | Aspherical Intraocular Lens
Number analyzed (Participants) | 20 | 20
μm | 0.10 (0.04) | 0.11 (0.04)

3. Secondary Outcome: Total Ocular High-order Aberrations
Description: A Hartmann-Shack aberrometer (Zywave, Bausch & Lomb Inc., Rochester, New York ) was used for measurement of HOAs of the whole eye. The measurements were done under maximal mydriasis with Mydrin-P (phenylephrine hydrochloride 0.5% and tropicamide 0.5%, Santen). The wavefront errors were described using the RMS of Zernike polynomials for total HOA at pupil diameters of 5 mm and 6 mm, primary spherical (Z 4,0) and 3rd-to 5th-order aberration at the pupil diameter of 6 mm.
Time Frame: average data of post-op 3rd, 6th, 12th week measurements
Measure: Mean (Standard Deviation); unit: μm
Groups:
- Aspherical Intraocular Lens: patients recieved cataract surgery and recived spherical intraocuar lens(Tecnis Z9000, AMO) in the other eye.
Arm/Group | Spherical Intraocular Lens | Aspherical Intraocular Lens
Number analyzed (Participants) | 20 | 20
μm | 0.6314 (0.1342) | 0.0856 (0.1070)

4. Primary Outcome: Best Corrected Contrast Sensitivity in Photopic Condition
Description: Contrast sensitivity testing was measured with spectacle correction for the target distance of three meters using a wall-mounted FACT sine-wave grating chart with nine levels of contrast (Stereo Optical Inc.)and five spatial frequency targets (1.5, 3, 6, 12, 18 cycles per degree (cpd)) at 250 lux. The last correct grating seen for each spatial frequency is recorded and translated by the "EYEVIEW™ Functional Analysis Software" into a log contrast sensitivity unit. The outcomes were recorded as average of the three post-operative measurements.
  ( physiological range of contrast sensitivity: 1.5 cpd : 25~82.5 ; 3 cpd: 30~150 ; 6 cpd: 65 ~ 200 ; 12 cpd: 20 ~130 ; 18 cpd: 6.5 ~ 65 )
Time Frame: average data of post-operative 3rd week, 6th week, 12th week measurements
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Aspheric Intraocular Lens: patients recieved cataract surgery and recived spherical intraocuar lens(Tecnis Z9000,AMO) in the other eye.
Arm/Group | Spherical Intraocular Lens | Aspheric Intraocular Lens
Number analyzed (Participants) | 20 | 20
units on a scale
  1.5 cpd | 47.03 (13.48) | 55.90 (20.76)
  3 cpd | 82.64 (14.78) | 85.09 (21.76)
  6 cpd | 69.31 (34.02) | 72.41 (31.45)
  12 cpd | 23.47 (17.73) | 27.45 (22.68)
  18 cpd | 6.97 (3.99) | 6.34 (4.51)

ADVERSE EVENTS:
Arm/Group | Cataract Patients
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No